CLINICAL TRIAL: NCT01135615
Title: Sevelamer, FGF-23 and Endothelial Dysfunction in CKD
Brief Title: Sevelamer, FGF-23 and Endothelial Dysfunction in Chronic Kidney Disease (CKD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GATAFGF23Sevelamer
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2010-05

CONDITIONS: We Investigated the Relationship Between Plasma FGF23 Levels and Endothelial Dysfunction in a Sizable Series of Incident Stage 3-4 CKD Patients.
Keywords: FGF-23, endothelial dysfunction, sevelamer
MeSH Terms: interventions — Sevelamer; calcium acetate

ARMS (2):
- Sevelamer (Other)
  Interventions: Drug: Sevelamer; Drug: calcium acetate
- calcium acetate (Other)
  Interventions: Drug: calcium acetate

INTERVENTIONS:
Drug: Sevelamer — The starting dose for sevelamer was 1-2 capsules (800 mg) three times a day
  Arms: Sevelamer
Drug: calcium acetate — calcium acetate (1000 mg) 1 tablet three times a day

SUMMARY:
Vascular calcification and endothelial dysfunction (ED) contribute to the development of cardiovascular disease (CVD) in patients with chronic kidney disease (CKD). Sevelamer, a non-calcium based phosphate binder, has been shown to attenuate cardiovascular calcification in CKD patients while the exact mechanism has not been clarified.

This study was designed to investigate the effect of short-term sevelamer treatment on both serum FGF23 levels concentrations and ED seen in CKD patients.

The researchers investigated the relationship between plasma FGF23 levels and the forearm blood flow response to ischemia in the forearm in a sizable series of incident stage 3-4 CKD patients.

DETAILED DESCRIPTION:
CKD stage 4 patients older than 18 years of age and willing to participate to the study were screened. Those who had serum phosphorus > 5.5 mg/dl were evaluated for the study. Patients with diabetes mellitus, history of coronary artery disease, smokers and those taking statins or renin-angiotensin blockers were excluded because of the effect of these factors on endothelial dysfunction. Of 192 screened patients 100 met the study criteria and were included in this study. Thirty-seven healthy subjects were studied as controls. The ethical committee of Gulhane School of Medicine approved the study and written informed consent was obtained from all patients.

Study design:

This was a randomized study conducted from 2008 through 2010 in Gulhane School of Medicine. The Outpatient Clinic of Department of Nephrology is a tertiary referral center. At admission, most patients were untreated (including phosphate binders) or treated only with antihypertensive agents. After the first evaluation, patients receiving phosphate binders (n=17) underwent a 2-week washout period. Patients who developed a phosphate level >5.5 mg/dl during this period were included in the study. Patients were randomly assigned in 1:1 ratio to receive sevelamer (Renagel capsule) or calcium acetate (Phos Ex tablet). The treatment phase was 8 weeks. During the study period serum calcium and phosphorus concentration were measured every 2 weeks and the dose of phosphate binders were titrated to achieve a serum phosphorus concentration < 5.5 mg/dl. The starting dose for sevelamer was 1-2 capsules (800 mg) three times a day and for calcium acetate (1000 mg) 1 tablet three times a day. The medications were given with meal and the doses were increased as needed. Patients were not given calcitriol during the study period.

Fasting blood samples were taken before and after the study to measure serum creatinine, serum albumin, hs-CRP, insulin, 25 (OH) Vit D, iPTH, lipid profile and serum FGF-23 concentration. Additionally, flow-mediated dilatation (FMD) and Intima Media Thickness (IMT) were also evaluated before and after the study.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 4 patients
* Older than 18 years of age
* Non-diabetic
* Serum phosphorus > 5.5 mg/dl

Exclusion Criteria:

* Diabetes mellitus
* History of coronary artery disease
* Smokers
* Taking statins or renin-angiotensin blockers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-01; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane School of Medicine, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Yilmaz MI, Sonmez A, Saglam M, Yaman H, Kilic S, Eyileten T, Caglar K, Oguz Y, Vural A, Yenicesu M, Mallamaci F, Zoccali C. Comparison of calcium acetate and sevelamer on vascular function and fibroblast growth factor 23 in CKD patients: a randomized clinical trial. Am J Kidney Dis. 2012 Feb;59(2):177-85. doi: 10.1053/j.ajkd.2011.11.007. Epub 2011 Dec 2. PMID 22137672